CLINICAL TRIAL: NCT03394092
Title: Changes in Glycopeptides of Serum Immunoglobulin G in Patients With Acute Myocardial Infarction and the Relationships Between Its Change and Prognosis
Brief Title: Serum Concentration of lgG in Patient With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Dalian Institute of Chemical Physics, Chinese Academy of Sciences , Dalian (Unknown)
Responsible Party: Sponsor
Other Study IDs: LCKY2017-1
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
Keywords: immunoglobulin G
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI: The study population consists of 50 patients with ST-elevated acute myocardial infarction (STEMI) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded. Blood is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture to assess the quantitative changes of IgG glycosylation by HPLC-MRM at 0 , 3 and 7 days after admission.
  Interventions: Diagnostic Test: Quantitative measurements the changes of IgG glycosylation
- Control: 50 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are studied as control group.Quantitative changes of IgG glycosylation be measured only once on admission.
  Interventions: Diagnostic Test: Quantitative measurements the changes of IgG glycosylation

INTERVENTIONS:
Diagnostic Test: Quantitative measurements the changes of IgG glycosylation — Serum (50 each group) is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture.Blood is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture to assess the quantitative changes of IgG glycosylation by HPLC-MRM at 0 , 3 and 7 days after admission.

SUMMARY:
The aim of this study is to investigate the changes in glycopeptides of serum immunoglobulin G in patients with acute myocardial infarction and the relationships between its change and prognosis.

DETAILED DESCRIPTION:
Immunoglobin G (IgG), a highly abundant glycoprotein in serum, is known to participate in blood immune responses.It has been an increasing interest in the analysis of the abnormal glycosylation of human lgG in healthy and disease states, such as autoimmune diseases and cancer.However, there is few relevant studies about the changes in glycopeptides of serum immunoglobulin G in patients with acute myocardial infarction. This study was performed for the frst timeto assess the quantitative changes of serum IgG glycosylation in patients with acute myocardial infarction and the relationships between its change and prognosis.

ELIGIBILITY:
Inclusion Criteria:

- diagnosed as STEMI.

* with left ventricular ejection fraction（LVEF）>=45%
* written informed consents are obtained
* admitted within 24 hours after chest pain attacked

Exclusion Criteria:

* complicated with rheumatic heart disease, coronary arteritis, hypertrophic cardiomyopathy or dilated cardiomyopathy

  * complicated with malignant tumor,the immune system diseases, blood system diseases, recently (within 2 weeks) taking glucocorticoid drugs, the use of immunosuppressive agents and cerebral infarction
  * with acute or chronic infection, surgery or trauma in the last month
  * secondary hypertension, severe liver dysfunction,severe renal insufficiency
  * with abnormal thyroid function or allergy to iodine agent refusal to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 with ST-elevation myocardial infarction (STEMI) patients and 50 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are studied as Control group. They will all undergo coronary angiography.The diagnosis is made according to American Heart Association(AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, asthma, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Serum quantitative determination of lgG | 12 months
  Quantitative measurements the changes of serum IgG glycosylation by HPLC-MRM

SECONDARY OUTCOMES:
Relationship between the serum hs-CRP and the quantitative level of lgG glycopeptides in peripheral blood. | 12 months
  correlation between the serum hs-CRP and lgG
MACEs during 12-month follow-up | 12 months
  Association of quantitative level of lgG with prognosis
The changes of LVEF in two groups | 12 months
  Association of quantitative level of lgG with the changes of cardiac function

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shinkawa T, Nakamura K, Yamane N, Shoji-Hosaka E, Kanda Y, Sakurada M, Uchida K, Anazawa H, Satoh M, Yamasaki M, Hanai N, Shitara K. The absence of fucose but not the presence of galactose or bisecting N-acetylglucosamine of human IgG1 complex-type oligosaccharides shows the critical role of enhancing antibody-dependent cellular cytotoxicity. J Biol Chem. 2003 Jan 31;278(5):3466-73. doi: 10.1074/jbc.M210665200. Epub 2002 Nov 8. PMID 12427744
- [Background] Hodoniczky J, Zheng YZ, James DC. Control of recombinant monoclonal antibody effector functions by Fc N-glycan remodeling in vitro. Biotechnol Prog. 2005 Nov-Dec;21(6):1644-52. doi: 10.1021/bp050228w. PMID 16321047
- [Background] Ferrara C, Grau S, Jager C, Sondermann P, Brunker P, Waldhauer I, Hennig M, Ruf A, Rufer AC, Stihle M, Umana P, Benz J. Unique carbohydrate-carbohydrate interactions are required for high affinity binding between FcgammaRIII and antibodies lacking core fucose. Proc Natl Acad Sci U S A. 2011 Aug 2;108(31):12669-74. doi: 10.1073/pnas.1108455108. Epub 2011 Jul 18. PMID 21768335
- [Background] Kaneko Y, Nimmerjahn F, Ravetch JV. Anti-inflammatory activity of immunoglobulin G resulting from Fc sialylation. Science. 2006 Aug 4;313(5787):670-3. doi: 10.1126/science.1129594. PMID 16888140
- [Background] Bruhns P, Samuelsson A, Pollard JW, Ravetch JV. Colony-stimulating factor-1-dependent macrophages are responsible for IVIG protection in antibody-induced autoimmune disease. Immunity. 2003 Apr;18(4):573-81. doi: 10.1016/s1074-7613(03)00080-3. PMID 12705859
- [Background] Quast I, Keller CW, Maurer MA, Giddens JP, Tackenberg B, Wang LX, Munz C, Nimmerjahn F, Dalakas MC, Lunemann JD. Sialylation of IgG Fc domain impairs complement-dependent cytotoxicity. J Clin Invest. 2015 Nov 2;125(11):4160-70. doi: 10.1172/JCI82695. Epub 2015 Oct 5. PMID 26436649
- [Background] Zou G, Ochiai H, Huang W, Yang Q, Li C, Wang LX. Chemoenzymatic synthesis and Fcgamma receptor binding of homogeneous glycoforms of antibody Fc domain. Presence of a bisecting sugar moiety enhances the affinity of Fc to FcgammaIIIa receptor. J Am Chem Soc. 2011 Nov 23;133(46):18975-91. doi: 10.1021/ja208390n. Epub 2011 Nov 1. PMID 22004528
- [Background] Everett BM, Pradhan AD, Solomon DH, Paynter N, Macfadyen J, Zaharris E, Gupta M, Clearfield M, Libby P, Hasan AA, Glynn RJ, Ridker PM. Rationale and design of the Cardiovascular Inflammation Reduction Trial: a test of the inflammatory hypothesis of atherothrombosis. Am Heart J. 2013 Aug;166(2):199-207.e15. doi: 10.1016/j.ahj.2013.03.018. Epub 2013 May 3. PMID 23895801
- [Background] Gala FA, Morrison SL. V region carbohydrate and antibody expression. J Immunol. 2004 May 1;172(9):5489-94. doi: 10.4049/jimmunol.172.9.5489. PMID 15100290
- [Background] Bondt A, Rombouts Y, Selman MH, Hensbergen PJ, Reiding KR, Hazes JM, Dolhain RJ, Wuhrer M. Immunoglobulin G (IgG) Fab glycosylation analysis using a new mass spectrometric high-throughput profiling method reveals pregnancy-associated changes. Mol Cell Proteomics. 2014 Nov;13(11):3029-39. doi: 10.1074/mcp.M114.039537. Epub 2014 Jul 8. PMID 25004930
- [Background] Plomp R, Dekkers G, Rombouts Y, Visser R, Koeleman CA, Kammeijer GS, Jansen BC, Rispens T, Hensbergen PJ, Vidarsson G, Wuhrer M. Hinge-Region O-Glycosylation of Human Immunoglobulin G3 (IgG3). Mol Cell Proteomics. 2015 May;14(5):1373-84. doi: 10.1074/mcp.M114.047381. Epub 2015 Mar 10. PMID 25759508
- [Background] Harre U, Lang SC, Pfeifle R, Rombouts Y, Fruhbeisser S, Amara K, Bang H, Lux A, Koeleman CA, Baum W, Dietel K, Grohn F, Malmstrom V, Klareskog L, Kronke G, Kocijan R, Nimmerjahn F, Toes RE, Herrmann M, Scherer HU, Schett G. Glycosylation of immunoglobulin G determines osteoclast differentiation and bone loss. Nat Commun. 2015 Mar 31;6:6651. doi: 10.1038/ncomms7651. PMID 25825024
- [Background] Moore JS, Wu X, Kulhavy R, Tomana M, Novak J, Moldoveanu Z, Brown R, Goepfert PA, Mestecky J. Increased levels of galactose-deficient IgG in sera of HIV-1-infected individuals. AIDS. 2005 Mar 4;19(4):381-9. doi: 10.1097/01.aids.0000161767.21405.68. PMID 15750391
- [Background] Russell AC, Simurina M, Garcia MT, Novokmet M, Wang Y, Rudan I, Campbell H, Lauc G, Thomas MG, Wang W. The N-glycosylation of immunoglobulin G as a novel biomarker of Parkinson's disease. Glycobiology. 2017 May 1;27(5):501-510. doi: 10.1093/glycob/cwx022. PMID 28334832
- [Background] Saldova R, Royle L, Radcliffe CM, Abd Hamid UM, Evans R, Arnold JN, Banks RE, Hutson R, Harvey DJ, Antrobus R, Petrescu SM, Dwek RA, Rudd PM. Ovarian cancer is associated with changes in glycosylation in both acute-phase proteins and IgG. Glycobiology. 2007 Dec;17(12):1344-56. doi: 10.1093/glycob/cwm100. Epub 2007 Sep 20. PMID 17884841
- [Background] Kazuno S, Furukawa J, Shinohara Y, Murayama K, Fujime M, Ueno T, Fujimura T. Glycosylation status of serum immunoglobulin G in patients with prostate diseases. Cancer Med. 2016 Jun;5(6):1137-46. doi: 10.1002/cam4.662. Epub 2016 Feb 16. PMID 26880719
- [Background] Yi CH, Weng HL, Zhou FG, Fang M, Ji J, Cheng C, Wang H, Liebe R, Dooley S, Gao CF. Elevated core-fucosylated IgG is a new marker for hepatitis B virus-related hepatocellular carcinoma. Oncoimmunology. 2015 Jul 7;4(12):e1011503. doi: 10.1080/2162402X.2015.1011503. eCollection 2015 Dec. PMID 26587313
- [Background] Hong Q, Lebrilla CB, Miyamoto S, Ruhaak LR. Absolute quantitation of immunoglobulin G and its glycoforms using multiple reaction monitoring. Anal Chem. 2013 Sep 17;85(18):8585-93. doi: 10.1021/ac4009995. Epub 2013 Aug 30. PMID 23944609
- [Background] Yang N, Goonatilleke E, Park D, Song T, Fan G, Lebrilla CB. Quantitation of Site-Specific Glycosylation in Manufactured Recombinant Monoclonal Antibody Drugs. Anal Chem. 2016 Jul 19;88(14):7091-100. doi: 10.1021/acs.analchem.6b00963. Epub 2016 Jun 24. PMID 27311011